CLINICAL TRIAL: NCT01327612
Title: A Phase 2 Open Label Extension Study of Conatumumab and AMG 479
Brief Title: Open Label Extension Study of Conatumumab and Ganitumab (AMG 479)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20101116; 2010-022270-14 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-04-01 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Advanced Solid Tumors; Carcinoid; Colorectal Cancer; Locally Advanced; Lymphoma; Metastatic Cancer; Non-Small Cell Lung Cancer; Sarcoma; Solid Tumors
Keywords: AMG 655; AMG 479; Apoptosis; Monoclonal Antibody; Tumor Necrosis Factor; Insulin-like Growth Factor; Bevacizumab; Modified FOLFOX6; mFOLFOX6; FOLFOX; Lymphoma; Trail Receptor; ganitumab; conatumumab
MeSH Terms: conditions — Carcinoid Tumor; Colorectal Neoplasms; Lymphoma; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Sarcoma | interventions — conatumumab; ganitumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Conatumumab Monotherapy (Experimental): Participants will continue to receive conatumumab every 2 weeks (Q2W) or every 3 weeks (Q3W) at the same dose and regimen as at the conclusion of the parent study.
  Interventions: Biological: Conatumumab
- Conatumumab + Ganitumab (Experimental): Participants will receive conatumumab and ganitumab by intravenous infusion at the same dose and regimen as at the conclusion of the parent study.
  Interventions: Biological: Conatumumab; Biological: Ganitumab
- Ganitumab Monotherapy (Experimental): Participants will continue to receive ganitumab Q3W or every 4 weeks (Q4W) at the same dose and regimen as at the conclusion of the parent study.
  Interventions: Biological: Ganitumab
- Conatumumab + mFOLFOX6 ± Bevacizumab (Experimental): Participants will continue to receive conatumumab by intravenous infusion in addition to modified FOLFOX6 chemotherapy with or without bevacizumab.
  Interventions: Drug: Modified FOLFOX6; Biological: Conatumumab; Biological: Bevacizumab

INTERVENTIONS:
Drug: Modified FOLFOX6 — The mFOLFOX6 regimen is a combination therapy of oxaliplatin 85 mg/m² administered as a 2-hour intravenous (IV) infusion on day 1 and leucovorin 400 mg/m² racemate or 200 mg/m² levo-leucovorin administered as a 2-hour infusion on day 1, followed by a loading dose of 5-fluorouracil (5-FU) 400 mg/m² IV bolus administered on day 1, then 5-FU 2400 mg/m² via ambulatory pump administered for a period of 46 to 48 hours every 14 days.
  Other Names: Oxaliplatin-Leucovorin-Fluorouracil chemotherapy
  Arms: Conatumumab + mFOLFOX6 ± Bevacizumab
Biological: Conatumumab — Administered by intravenous infusion Q2W or Q3W.
  Other Names: AMG 655
  Arms: Conatumumab + Ganitumab; Conatumumab + mFOLFOX6 ± Bevacizumab; Conatumumab Monotherapy
Biological: Ganitumab — Administered by intravenous infusion Q3W or Q4W.
  Other Names: AMG 479
  Arms: Conatumumab + Ganitumab; Ganitumab Monotherapy
Biological: Bevacizumab — Administered at a dose of 5 mg/kg by intravenous infusion on day 1 of each 14 day cycle.
  Other Names: Avastin
  Arms: Conatumumab + mFOLFOX6 ± Bevacizumab

SUMMARY:
The purpose of this protocol is to allow continued treatment with conatumumab and/or ganitumab, with or without chemotherapy, to participants who completed a separate Amgen-sponsored conatumumab or ganitumab study without disease progression whose previous studies were closed.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in this study, subjects must be currently enrolled in a prior Amgen-sponsored conatumumab or AMG 479 study and are eligible according to the parent study to receive their next dose of conatumumab (with or without co-therapy), or AMG 479 alone.

Subjects must have their eligibility assessed for this study and be enrolled within 30 days of their last treatment on the parent protocol

Exclusion Criteria:

* Discontinued from a conatumumab study due to an adverse event considered by the investigator to be related to conatumumab treatment, including intolerance to conatumumab
* Subjects determined to have disease progression during their participation in the parent Amgen study
* Woman or man with partner of childbearing potential not consenting to use adequate contraceptive precautions ie, double barrier contraceptive methods (eg, diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last dose of protocol-specified therapy administration
* Subject is pregnant or breast feeding, or planning to become pregnant within 6 months after the last dose of protocol-specified therapy administration
* Male subject with a pregnant partner who is not willing to use a condom during treatment and for an additional 6 months after the last dose of protocol-specified therapy administration
* Subject has previously entered this study
* Subject will not be available for protocol required study visits, to the best of the subject and investigator's knowledge
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (10):
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Denver, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Ann Arbor, Michigan
  - Research Site, Buffalo, New York
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Ogden, Utah
- Research Site, Szczecin, Poland
- Research Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants with different types of solid tumors who had completed one of the following Amgen-sponsored conatumumab or ganitumab studies:
  20050118 (NCT00562380) 20050171 20060295 (NCT00534027) 20060340 (NCT00791011) 20060464 (NCT00625651) 20070411 (NCT00819169). Participants who had not progressed in the parent study were eligible to participate in this trial.
  The study was conducted at 12 centers in the United States, Spain, and Poland.
Pre-assignment Details: This was an extension study that permitted participants to continue treatment with conatumumab, with or without co-therapy (modified FOLFOX6 chemotherapy with or without bevacizumab, or ganitumab), or with ganitumab alone, administered at the same dose level and schedule that participants received at the conclusion of the parent study. Participants remained on treatment until disease progression, intolerability, or withdrawal of consent.
  Results are reported by parent study and treatment.
Groups:
- 20050118: Ganitumab 20 mg/kg: Ganitumab 20 mg/kg once every 4 weeks by intravenous infusion.
- 20050171: Conatumumab 0.45 mg/kg: Conatumumab 0.45 mg/kg every 2 weeks by intravenous infusion.
- 20060295: Conatumumab 3 mg/kg: Conatumumab 3 mg/kg every 3 weeks by intravenous infusion.
- 20060340: Conatumumab 5 mg/kg: Conatumumab 5 mg/kg once every 3 weeks by intravenous infusion.
- 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab: Conatumumab 2 mg/kg once every 2 weeks by intravenous infusion in addition to modified FOLFOX6 (mFOLFOX6) chemotherapy and bevacizumab 5 mg/kg once every 2 weeks.
- 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab: Conatumumab 10 mg/kg once every 2 weeks by intravenous infusion in addition to modified FOLFOX6 chemotherapy, with or without bevacizumab 5 mg/kg once every 2 weeks.
- 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg: Conatumumab 15 mg/kg + ganitumab 18 mg/kg once every 3 weeks by intravenous infusion.
Period: Overall Study
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Started | 2 | 1 | 1 | 1 | 2 | 3 | 2
Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 1 | 1 | 1 | 0 | 1 | 2 | 2
Not completed — Administrative Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of conatumumab or ganitumab.
Groups:
- 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab: Conatumumab 2 mg/kg once every 2 weeks by intravenous infusion in addition to modified FOLFOX6 chemotherapy and bevacizumab 5 mg/kg once every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg | Total
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (14.1) | 57.0 | 44.0 | 46.0 | 66.5 (7.8) | 56.3 (8.7) | 68.0 (15.6) | 58.8 (11.1)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 8
  65 - 74 years | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  75 - 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ≥ 85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 5
  Male | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 1 | 1 | 2 | 3 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a clinical trial participant, including worsening of a pre-existing medical condition. The event does not necessarily have a causal relationship with study treatment.
Time Frame: From first dose of study drug in the extension study to 30 days after last dose; median duration of treatment with conatumumab was 1190.5 days and 1163.0 days for ganitumab.
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Count of Participants; unit: Participants
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
Participants | 2 | 1 | 1 | 1 | 2 | 3 | 2

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event is defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal,
  * life threatening (places the participant at immediate risk of death),
  * required in-patient hospitalization or prolongation of existing hospitalization,
  * resulted in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other medically important serious event.
Time Frame: as for outcome 1
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Count of Participants; unit: Participants
Groups:
- 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg: Conatumumab 15 mg/kg and ganitumab 18 mg/kg once every 3 weeks by intravenous infusion.
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
Participants | 1 | 0 | 1 | 0 | 1 | 3 | 2

3. Secondary Outcome: Maximum Change From Baseline in Blood Pressure
Description: Maximum change from baseline is defined for each participant as the maximum change from baseline value observed across all visits.
Time Frame: Baseline and day 1 of each treatment cycle (every 2, 3, or 4 weeks depending on dosing schedule) up to 30 days after last dose; median duration of treatment with conatumumab was 1190.5 days and 1163.0 days for ganitumab.
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
mmHg
  Systolic blood pressure | 5.5 (9.2) | 7.0 | 54.0 | 37.0 | 42.0 (0.0) | 26.0 (17.3) | 32.5 (31.8)
  Diastolic blood pressure | 7.5 (9.2) | 1.0 | 10.0 | 13.0 | 27.5 (9.2) | 14.7 (6.4) | 23.5 (6.4)

4. Secondary Outcome: Minimum Change From Baseline in Blood Pressure
Description: Minimum change from baseline is defined for each participant as the minimum change from baseline value observed across all visits.
Time Frame: as for outcome 3
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
mmHg
  Systolic blood pressure | -28.5 (17.7) | -45.0 | -20.0 | -21.0 | -22.5 (16.3) | -29.0 (10.8) | -12.0 (12.)
  Diastolic blood pressure | -19.5 (9.2) | -27.0 | -20.0 | -25.0 | -8.5 (7.8) | -14.3 (5.5) | -10.0 (4.2)

5. Secondary Outcome: Number of Participants With CTCAE Grade 3 or Higher Clinical Laboratory Toxicities
Description: Laboratory toxicities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: as for outcome 1
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Count of Participants; unit: Participants
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
Participants | 0 | 0 | 1 | 0 | 2 | 2 | 1

6. Secondary Outcome: Best Overall Response
Description: Radiological assessments to evaluate disease extent (with change compared to nadir from the parent protocol) were performed at regular intervals, at a minimum once every 6 months or more frequently if clinically indicated (starting from their last scan on the parent protocol), per standard of care (SOC) at each facility. Tumor response was assessed by the Investigator as either complete response, partial response, stable disease, or progressive disease.
Time Frame: Approximately every 6 months until end of treatment; median duration of treatment with conatumumab was 1190.5 days and 1163.0 days for ganitumab.
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Count of Participants; unit: Participants
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
Participants
  Complete response | 0 | 1 | 0 | 1 | 1 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Stable disease | 2 | 0 | 1 | 0 | 0 | 2 | 1
  Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Disease Progression or Death Due to Disease Progression
Time Frame: as for outcome 1
Population: Participants who received at least one dose of conatumumab or ganitumab.
Measure: Count of Participants; unit: Participants
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 1 | 2 | 3 | 2
Participants
  Disease progression | 1 | 1 | 1 | 0 | 2 | 2 | 2
  Death due to disease progression | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug in the extension study to 30 days after last dose; median duration of treatment with conatumumab was 1190.5 days and 1163.0 days for ganitumab.
Arm/Group | 20050118: Ganitumab 20 mg/kg | 20050171: Conatumumab 0.45 mg/kg | 20060295: Conatumumab 3 mg/kg | 20060340: Conatumumab 5 mg/kg | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/1 | 1/2 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 1/1 | 0/1 | 1/2 | 3/3 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 1/1 | 2/2 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20050118: Ganitumab 20 mg/kg (N=2) | 20050171: Conatumumab 0.45 mg/kg (N=1) | 20060295: Conatumumab 3 mg/kg (N=1) | 20060340: Conatumumab 5 mg/kg (N=1) | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab (N=2) | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab (N=3) | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg (N=2)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transurethral bladder resection (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20050118: Ganitumab 20 mg/kg (N=2) | 20050171: Conatumumab 0.45 mg/kg (N=1) | 20060295: Conatumumab 3 mg/kg (N=1) | 20060340: Conatumumab 5 mg/kg (N=1) | 20060464: Conatumumab 2 mg/kg + mFOLFOX6 + Bevacizumab (N=2) | 20060464: Conatumumab 10 mg/kg + mFOLFOX6 ± Bevacizumab (N=3) | 20070411: Conatumumab 15 mg/kg + Ganitumab 18 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Micrographic skin surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin neoplasm excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
May-Thurner syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT01327612/Prot_000.pdf
  • Statistical Analysis Plan (2010-12-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT01327612/SAP_001.pdf